CLINICAL TRIAL: NCT03924843
Title: Responsivity and Reproducibility of Messenger and Micro RNA Airway Inflammatory Markers - a Pilot Study
Brief Title: mRNA and miRNA Airway Inflammatory Markers
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Huib A.M. Kerstjens, Full professor pulmonology; Head of department of Pulmonology and Tuberculosis; Principal Investigator, University Medical Center Groningen
Other Study IDs: NL 62038.042.17
Record Dates: First submitted 2019-03-06; First posted 2019-04-23 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: COPD; COPD Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Induced sputum samples; nasal mucosa samples
  Main study parameters:
  * mRNA level expression of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta
  * miRNA level expression of IL-6, IL-8, IL-17, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta
  * inflammatory cell profiles, LTB4 and protein levels of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta, ECP and TGF-beta
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates cytokine Messenger (mRNA) and microRNA (miRNA) level expression of interleukin (IL) -6, IL-8, IL-17, tumor necrosis factor (TNF)-alpha, monocyte chemoattractant protein (MCP)-1, macrophage inflammatory protein (MIP)-1 beta and transforming growth factor (TGF)-beta regarding their reproducibility and responsivity in induced sputum and nasal mucosa of patients with chronic obstructive pulmonary disease (COPD) in order to assess their potential as a biomarker outcome measure.

DETAILED DESCRIPTION:
Rationale:There is an increased interest to identify sensitive airway biomarkers in order to evaluate the potential and efficacy of anti-inflammatory and -remodelling therapeutic interventions. Biomarkers should be easily obtainable, reliable and valid. In COPD, easily obtainable would suggest use of blood, or more directly associated with the airways: sputum or epithelial brushes. Sputum is an obvious opportunity. It has been shown that gene expression changes in the nasal mucosa might be used as suitable surrogate for epithelial cells of the lower airways in patients with airway inflammatory diseases. However, further studies are needed to validate these assumptions. Measurement of messenger RNA, and of micro RNA derived from sputum samples and nasal brushes would fulfil the ease of use required of a biomarker. Messenger RNA would allow for easier quantification in variable dilution samples (sputum). The Groningen Research Institute for Asthma and COPD (GRIAC research group) has experience with sputum and nasal brushes, mRNA and miRNA, but more information is needed on especially reproducibility of the measurements, as well as on responsivity. Both are a prerequisite when designing new intervention trials with such biomarkers.

Therefore, the aim of this study is to investigate cytokine messenger and microRNA level expression of IL-6, IL-8, IL-17, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta regarding their reproducibility and responsivity in induced sputum and nasal mucosa of COPD patients in order to assess their potential as an objective outcome measure.

The primary objectives of this prospective pilot study are the determination of the reproducibility and responsivity of mRNA level expression of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta, ECP and TGF-beta as airway inflammatory markers in induced sputum as well as mRNA and miRNA expression levels of IL-6, IL-8, IL-17, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta as airway inflammatory markers in nasal mucosa. The secondary objective includes the analyses of the measurement characteristics of inflammation cell profiles, LTB4 and protein levels of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta, ECP and TGF-beta.

Twenty COPD patients with an initial COPD exacerbation will be followed for a period of seven weeks for three consecutive visits

The main parameters of induced sputum samples will be mRNA level expression of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta. The main parameters of nasal mucosa samples will be mRNA and miRNA level expression of IL-6, IL-8, IL-17, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta.

To allow for full perspective on the outcomes, inflammatory cell profiles, Leukotriene B4 (LTB4) and protein levels of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta, eosinophilic cationic protein (ECP) and TGF-beta in sputum will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men/Women age >40 years.
* Diagnoses of COPD according to criteria of the American Thoracic Society (ATS), a disease state characterized by the presence of chronic airway obstruction due to chronic bronchitis (cough/sputum on most days a week for 3 months in a year for at least two successive years) and/or emphysema
* Diagnosis of moderate or severe COPD exacerbation (see "Definitions")
* FEV1 > 0.8 L and ability to produce sputum after hypertonic saline production
* Post bronchodilator FEV1/Forced Vital Capacity (FVC) ratio <70 % and post bronchodilator FEV1< 80% pred.
* A smoking history of >10 pack years

Exclusion Criteria:

* Pneumonia as determined by X-ray
* > 48 h intake of prednisolon/antibiotics
* Need for mechanical ventilation (either invasive or non-invasive)
* Treatment with immune-modulating agents for any disease
* Experimental interventions for COPD last half year
* Former/concomitant diagnosis of asthma
* Any significant other pulmonary disease or disorder
* Other significant disease or disorder (like alpha-1-antitrypsine deficiency, significant bronchiectasis, cardiovascular, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic (including diagnosed diabetes), malignant, psychiatric, major physical impairment), which, in the opinion of the investigators may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study.
* Existing pregnancy/ current willingness for becoming pregnant

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Twenty COPD patients with an initial COPD exacerbation will be followed for a period of seven weeks for three consecutive visits
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change of mRNA cytokine expression measured in induced sputum samples | Change of outcome measures will be assessed during one COPD exacerbation phase, after 42 days and after 44-51 days
  mRNA level expression of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta
Change of miRNA and mRNA cytokine expression measured in nose mucosa samples | Change of outcome measures will be assessed during one COPD exacerbation phase, after 42 days and after 44-51 days
  mRNA and miRNA level expression of IL-6, IL-8, IL-17, TNF-alpha, MCP-1, MIP-1 beta and TGF-beta

SECONDARY OUTCOMES:
Change of inflammatory cell profiles, LTB4 levels and protein cytokine levels measured in induced sputum samples | Change of outcome measures will be assessed during one COPD exacerbation phase, after 42 days and after 44-51 days
  Inflammatory cell profiles; LTB4 levels; protein levels of IL-6, IL-8, TNF-alpha, MCP-1, MIP-1 beta, ECP and TGF-beta

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center; Department of Pulmonary Diseases, Groningen, Netherlands

REFERENCES:
- [Background] Bathoorn E, Liesker J, Postma D, Koeter G, van Oosterhout AJ, Kerstjens HA. Safety of sputum induction during exacerbations of COPD. Chest. 2007 Feb;131(2):432-8. doi: 10.1378/chest.06-2216. PMID 17296644
- [Background] Brightling CE, Monterio W, Green RH, Parker D, Morgan MD, Wardlaw AJ, Pavord D. Induced sputum and other outcome measures in chronic obstructive pulmonary disease: safety and repeatability. Respir Med. 2001 Dec;95(12):999-1002. doi: 10.1053/rmed.2001.1195. PMID 11778799
- [Background] Comer DM, Elborn JS, Ennis M. Comparison of nasal and bronchial epithelial cells obtained from patients with COPD. PLoS One. 2012;7(3):e32924. doi: 10.1371/journal.pone.0032924. Epub 2012 Mar 6. PMID 22412951
- [Background] Hogg JC, Chu F, Utokaparch S, Woods R, Elliott WM, Buzatu L, Cherniack RM, Rogers RM, Sciurba FC, Coxson HO, Pare PD. The nature of small-airway obstruction in chronic obstructive pulmonary disease. N Engl J Med. 2004 Jun 24;350(26):2645-53. doi: 10.1056/NEJMoa032158. PMID 15215480
- [Background] Huang CC, Wang CH, Fu CH, Huang CC, Chang PH, Chen YW, Wu CC, Wu PW, Lee TJ. Association between cigarette smoking and interleukin-17A expression in nasal tissues of patients with chronic rhinosinusitis and asthma. Medicine (Baltimore). 2016 Nov;95(47):e5432. doi: 10.1097/MD.0000000000005432. PMID 27893686
- [Background] Kistemaker LE, Oenema TA, Meurs H, Gosens R. Regulation of airway inflammation and remodeling by muscarinic receptors: perspectives on anticholinergic therapy in asthma and COPD. Life Sci. 2012 Nov 27;91(21-22):1126-33. doi: 10.1016/j.lfs.2012.02.021. Epub 2012 Mar 3. PMID 22406302
- [Background] O'Donnell RA, Peebles C, Ward JA, Daraker A, Angco G, Broberg P, Pierrou S, Lund J, Holgate ST, Davies DE, Delany DJ, Wilson SJ, Djukanovic R. Relationship between peripheral airway dysfunction, airway obstruction, and neutrophilic inflammation in COPD. Thorax. 2004 Oct;59(10):837-42. doi: 10.1136/thx.2003.019349. PMID 15454648
- [Background] Perng DW, Tao CW, Su KC, Tsai CC, Liu LY, Lee YC. Anti-inflammatory effects of salmeterol/fluticasone, tiotropium/fluticasone or tiotropium in COPD. Eur Respir J. 2009 Apr;33(4):778-84. doi: 10.1183/09031936.00115308. Epub 2009 Jan 7. PMID 19129278
- [Background] Powrie DJ, Wilkinson TM, Donaldson GC, Jones P, Scrine K, Viel K, Kesten S, Wedzicha JA. Effect of tiotropium on sputum and serum inflammatory markers and exacerbations in COPD. Eur Respir J. 2007 Sep;30(3):472-8. doi: 10.1183/09031936.00023907. Epub 2007 May 15. PMID 17504798
- [Background] Rutgers SR, Postma DS, ten Hacken NH, Kauffman HF, van Der Mark TW, Koeter GH, Timens W. Ongoing airway inflammation in patients with COPD who Do not currently smoke. Chest. 2000 May;117(5 Suppl 1):262S. doi: 10.1378/chest.117.5_suppl_1.262s. No abstract available. PMID 10843943
- [Background] Singh D, Edwards L, Tal-Singer R, Rennard S. Sputum neutrophils as a biomarker in COPD: findings from the ECLIPSE study. Respir Res. 2010 Jun 15;11(1):77. doi: 10.1186/1465-9921-11-77. PMID 20550701
- [Background] Wessler I, Kirkpatrick CJ. Acetylcholine beyond neurons: the non-neuronal cholinergic system in humans. Br J Pharmacol. 2008 Aug;154(8):1558-71. doi: 10.1038/bjp.2008.185. Epub 2008 May 26. PMID 18500366
- [Background] Zhang X, Sebastiani P, Liu G, Schembri F, Zhang X, Dumas YM, Langer EM, Alekseyev Y, O'Connor GT, Brooks DR, Lenburg ME, Spira A. Similarities and differences between smoking-related gene expression in nasal and bronchial epithelium. Physiol Genomics. 2010 Mar 3;41(1):1-8. doi: 10.1152/physiolgenomics.00167.2009. Epub 2009 Dec 1. PMID 19952278